CLINICAL TRIAL: NCT01186926
Title: Australian Prospective Clinical Study of the Apnex Medical Hypoglossal Nerve Stimulation (HGNS) System to Treat Obstructive Sleep Apnea
Brief Title: Australian Clinical Study of the Apnex Medical HGNS System to Treat Obstructive Sleep Apnea
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Apnex Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-003
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2011-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; OSA; hypoglossal nerve stimulation; sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HGNS Treatment (Experimental)
  Interventions: Device: HGNS Treatment

INTERVENTIONS:
Device: HGNS Treatment — The Apnex Hypoglossal Nerve Stimulation (HGNS) System is an implanted medical device that is designed to prevent the tongue from blocking the airway during sleep. It is fully automatic and can be implanted during a simple surgical procedure. After it is implanted, the device is programmed to meet the unique needs of each patient. The device is on when the patient is sleeping, and off when the patient is awake.

SUMMARY:
The overall goal of the study is to evaluate the safety, efficacy and therapy settings of the HGNS System for stimulating the hypoglossal nerve to help maintain an open airway in subjects with obstructive sleep apnea (OSA).

ELIGIBILITY:
Eligibility Criteria

1. Previously diagnosed with moderate to severe obstructive sleep apnea.
2. Subject has failed or does not tolerate CPAP treatment.
3. Age between 21 and 70 years.
4. Body mass index (BMI) less than or equal to 40

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Mean change in AHI measured with in-lab nighttime polysomnography (PSG) compared to baseline | 6 months post-implant
Adverse event profile interoperatively, perioperatively, and long term post implant | 1, 3, 6, 12, 24, and 36 months post implant

SECONDARY OUTCOMES:
Mean change in functional outcomes measured with the Functional Outcomes of Sleep Questionnaire (FOSQ) compared to baseline | 6 months post-implant

CONTACTS AND LOCATIONS:
Overall Officials: Maree Barnes, MD, Principal Investigator — Institute for Breathing and Sleep, Austin Health; David Hillman, MD, Principal Investigator — West Australian Sleep Disorders Research Institute, St. Charles Gardner Hospital; Doug McEvoy, MD, Principal Investigator — Adelaide Institute for Sleep Health, Repatriation General Hospital; John Wheatley, MD, Principal Investigator — Westmead Hospital Dept of Respiratory Medicine

REFERENCES:
- [Result] Eastwood PR, Barnes M, Walsh JH, Maddison KJ, Hee G, Schwartz AR, Smith PL, Malhotra A, McEvoy RD, Wheatley JR, O'Donoghue FJ, Rochford PD, Churchward T, Campbell MC, Palme CE, Robinson S, Goding GS, Eckert DJ, Jordan AS, Catcheside PG, Tyler L, Antic NA, Worsnop CJ, Kezirian EJ, Hillman DR. Treating obstructive sleep apnea with hypoglossal nerve stimulation. Sleep. 2011 Nov 1;34(11):1479-86. doi: 10.5665/sleep.1380. PMID 22043118
- See also: Related Info — http://www.apnexmedical.com